CLINICAL TRIAL: NCT01928134
Title: The Efficacy of Vitamin K2 on Human Osteoporosis, Blood-vessel Calcification and Sclerosis
Brief Title: The Efficacy of Vitamin K2 n Human Osteoporosis, Blood-vessel Calcification and Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Shih-Li Su, Attending Physician of Section of Endocrinology and Metabolism, Changhua Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VitK2
Record Dates: First submitted 2013-08-19; First posted 2013-08-23 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: Vitamin K2; Vitamin D3; Bioavailability of calcium; volunteers; Men; non-pregnant women; twenty years of age
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Vit K2+ Vit D3+ calcium carbonate (CaCO3)
  Interventions: Dietary Supplement: Vit K2+ Vit D3+ calcium carbonate (CaCO3)
- B (Active Comparator): Vit K2+CaCO3
  Interventions: Dietary Supplement: Vit K2+CaCO3

INTERVENTIONS:
Dietary Supplement: Vit K2+ Vit D3+ calcium carbonate (CaCO3)
  Arms: A
Dietary Supplement: Vit K2+CaCO3
  Arms: B

SUMMARY:
This study used the generally recognized as safe (GRAS) grade of Bacillus subtilis natto to produce Vitamin K2, Menaquinone-7(MK-7), via fermentation, for functional evaluation. There are four major objectives for this study: (1) bioavailability of calcium; (2) evaluation of bone density improvement; (3) evaluation of blood-vessel calcification and sclerosis improvement; (4) safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Men and non-pregnant women who are at least 20 years and under 75 years of age; and
2. Female subjects cannot be pregnant or breast feeding.
3. Patients who are, in the opinion of the Investigator, able to comply with the requirements of the study; and
4. Patients who have been adequately informed of the nature and risks of the study and who have given written informed consent prior to receiving study medication.

Exclusion Criteria:

1. Women who are pregnant, as determined by a urine pregnancy test, or breast-feeding.
2. Presence or history of congestive heart failure (NYHA class III/IV) within the prior 12 weeks.
3. Recent myocardial infarction (within the prior 12 weeks).
4. Unstable angina pectoris.
5. Known or suspected renal insufficiency defined as creatinine>1.5mg/dl.
6. Known or suspected hepatic insufficiency defined as abnormal liver function tests (GOT/GPT) >3x upper normal limit (i.e., 120 U/l).
7. Known hypomotility syndrome: (such as hypothyroidism or scleroderma).
8. Recent major trauma within the prior 12 weeks.
9. Recent surgery requiring anesthesia including coronary artery bypass graft (within 12 weeks).
10. Recent hospitalization (within 12 weeks)
11. Uncontrolled hypertension (defined as a systolic blood pressure>180mmHg or a diastolic blood pressure >105mmHg).
12. Uncontrolled hyperlipidemia (defined as total cholesterol>240mg/dL or triglyceride >200mg/dL).
13. Uncontrolled diabetes (defined as HbA1c>7%).
14. Cigarette smoker (>=1/day).
15. Acute infection requiring current antibiotic therapy.
16. Current use of anticoagulant medication (e.g., warfarin).
17. Recent or abrupt change (within 1 month) in usual diet.
18. Use of an investigational drug (within 30 days prior to enrollment).
19. Known allergies to the component of study medication
20. Patients have acute disease, and in the opinion of investigators, are not suitable to participate in this study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-04; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Serum Calcium | at 4 hours after intake

SECONDARY OUTCOMES:
Change from baseline in urine calcium/creatinine ratio | at 4 hours after intake

OTHER OUTCOMES:
Change from baseline in serum Parathyroid hormone(PTH) | at 4 hour after intake

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Li Su, MD, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan, Taiwan